CLINICAL TRIAL: NCT01563614
Title: Safety and Efficacy of Liposomal Cytarabine in Combination With Radiotherapy (RT) and Lomustine for the Treatment of Leptomeningeal Metastasis From Malignant Melanoma
Brief Title: A Clinical Trial to Assess the Safety & Efficacy of the Treatment of Patients With Metastasis From Malignant Melanoma - Treatment Consists of the Substances Lomustine (Capsules) & Cytarabine (Injected Into an Area Near the Spinal Cord), Accompanied by Radiotherapy of the Brain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients can be recruited for this trial anymore due to other therapeutical approaches that became available.
Sponsor: University Hospital, Bonn (Other)
Collaborators: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Principal Investigator, PD Dr. Martin Glas, Deputy Director Division of Clinical Neurooncology Unit, University Hospital, Bonn
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DepoRaCe
Record Dates: First submitted 2012-03-09; First posted 2012-03-27 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Leptomeningeal Metastasis From Malignant Melanoma
MeSH Terms: interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Brain radiotherapy concomitant to lomustine and liposomal cytarabine chemotherapy.
  Interventions: Radiation: Brain radiotherapy (WBRT alone, SRT/SRS alone or WBRT plus SRT/SRS); Drug: Lomustine; Drug: Liposomal cytarabine

INTERVENTIONS:
Radiation: Brain radiotherapy (WBRT alone, SRT/SRS alone or WBRT plus SRT/SRS) — Brain radiotherapy concomitant to lomustine and liposomal cytarabine chemotherapy.
Drug: Lomustine — Brain radiotherapy concomitant to lomustine and liposomal cytarabine chemotherapy.
Drug: Liposomal cytarabine — Brain radiotherapy concomitant to lomustine and liposomal cytarabine chemotherapy.

SUMMARY:
The purpose of this trial is to test the safety and tolerance of the combination therapy with cytarabine, lomustine and radiotherapy in patients with leptomeningeal metastasis from malignant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Malignant melanoma (including melanoma of unknown primary site, recurrent and pretreated systemic melanoma and/or melanoma with parenchymal CNS metastases) with leptomeningeal metastasis as demonstrated by a positive CSF (cerebrospinal liquor) cytology AND/OR by the presence of characteristic signs and symptoms of leptomeningeal metastasis supported by an MRI scan indicating the presence of meningeal tumour
* CSF flow abnormalities must be excluded
* Males or females ≥ 18 years of age
* Karnofsky Performance Status > 50%
* Adequate organ function (adequate bone marrow reserve, adequate liver function, adequate renal function. adequate blood clotting)

Exclusion Criteria:

* Unresected parenchymal brain metastases with a diameter > 3 cm
* Prior non melanoma malignancy (unless adequately treated carcinoma in situ of the cervix or non melanoma skin cancer)
* Prior intrathecal chemotherapy
* Prior treatment with systemic cytarabine or nitrosureas
* The patient ist pregnant or breast feeding
* Severe, active co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerance | 30 weeks
  The primary endpoint is safety and tolerance and will be based on the frequency and severity of adverse events.

SECONDARY OUTCOMES:
Delay of treatments | 30 weeks
  Frequency and median time of delay of each of the treatments (lomustine, liposomal cytarabine, radiotherapy).
Response rate | 30 weeks
  Overall response rate determined by clinical, MRI- and CSF-cytological assessment criteria.
Progression | 30 weeks
  Neurological progression, progression free survival, overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Glas, PD Dr., Principal Investigator — Neurologische Universitaetsklinik Bonn
Locations (1):
- Neurologische Universitaetsklinik Bonn, Bonn, Germany